CLINICAL TRIAL: NCT02657304
Title: Effect of Early Education and Information of Sleep Apnea on the Observance of CPAP Treatment
Brief Title: Effect of Early Education on the Observance of CPAP Treatment
Acronym: CoachSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1508146; 2015-A01635-44 (Other: ANSM)
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Sleep Apnea Syndrome
Keywords: Sleep Apnea; CPAP
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coaching group (Experimental): PPC + Coaching
  Interventions: Behavioral: Coaching group
- Control group (Active Comparator): PPC
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Coaching group — patients will have a medical consultation at 2 weeks post-diagnostic and one phone call/month for duration of 5 months. The consultations will use visual support, CPAP device and its accessories.
  Arms: Coaching group
Other: Control group — patients receive only usual care (standard), it's mean: diagnosis with explanation of the disease and benefit of CPAP, entrusts a medical device provider, then an appointment proposed by the doctor or taken by the patient (5 months).
  Arms: Control group

SUMMARY:
Sleep apnea (SA) affects more than 4% from general population and is largely underdiagnosed. SA can increase the occurrence of cardiovascular, endocrine and metabolic events (particularly stroke, diabetes & obesity). CPAP is currently the Gold Standard treatment of SA and to prevent these events, with a major clinical benefit, long term adherence to CPAP is a significant problem where a significant rate of rejection and abundance after 6 months of treatment.

DETAILED DESCRIPTION:
Sleep apnea (SA) affects more than 4% from general population (20% of people over 65 years) and is largely underdiagnosed, it can be rise up by some factors such as: obesity, male gender. Sleep Apnea can increase the occurrence of cardiovascular, endocrine and metabolic events (particularly stroke, diabetes & obesity). CPAP is currently the Gold Standard treatment of SA and to prevent these events, with a major clinical benefit, long term adherence to CPAP is a significant problem where a significant rate of rejection and abundance after 6 months of treatment.

The investigators hypothesize that an early education and information of SA (in the first 2 weeks after diagnosis of SA and one telephonic call/month while 5 months) would allow to increase significantly the optimal observance of CPAP (> 5 h/night).

Thus, in this study, we will compare evolution of the observance of CPAP (h/night), of the apnea hypopnea index (AHI), patient knowledge of their SA and its deleterious health consequences in an early education and information during five months against a control group receiving only usual care (standard).

ELIGIBILITY:
Inclusion Criteria:

* Patients affiliated or entitled to a French medical insurance
* Patients of both gender, aged from 18 to 80 years
* Patients with AHI > 30/hour or between 15 & 30/h with Sleep Fragmentation Index (SFI) of more than 10/h
* Signature of consent

Exclusion Criteria:

* Known diseases which contraindicated used of CPAP treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Observance | 5 months
  Percentage of patients with a mean duration of observance of more than 5h/night after five months of follow-up in the coached and the control groups

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No